CLINICAL TRIAL: NCT04127929
Title: 12-Month Clinical Performance Evaluation of a Current Glass Carbomer Restorative System
Brief Title: Investigation of Glass Carbomer Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Okan University (Other)
Collaborators: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Zeynep Buket Kaynar, Principal Investigator, Okan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 280486
Record Dates: First submitted 2019-10-04; First posted 2019-10-16 (Actual); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Dental Caries
Keywords: glass ionomer, composite, clinical
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Glass carbomer (Active Comparator)
  Interventions: Other: Restoration of cavities using glass carbomer material (GCP Dental)
- Tokuyama Estelite Posterior (Active Comparator)
  Interventions: Other: Restoration of cavities using nanocomposite resin (Tokuyama Estelite Posterior)

INTERVENTIONS:
Other: Restoration of cavities using glass carbomer material (GCP Dental) — Detection of caries then restoration of cavities
  Arms: Glass carbomer
Other: Restoration of cavities using nanocomposite resin (Tokuyama Estelite Posterior) — Detection of caries then restoration of cavities
  Arms: Tokuyama Estelite Posterior

SUMMARY:
The aim of this in vivo study was to evaluate the clinical 1 year follow-up of silica and flouroapatite reinforced glass carbomer filling material.

DETAILED DESCRIPTION:
The aim of this in vivo study was to evaluate the clinical 1 year follow-up of silica and flouroapatite reinforced glass carbomer filling material.

In this study, total of 100 (46 class I, 54 class II) restorations were performed in 36 patients. All cavities were prepared conventionally. Half of the restorations were restored with nano composite resin (Tokuyama Estelite, Tokuyama Dental, Japan) and the other half were restored with glass carbomer material (GCP Dental, The Netherlands). Rubber-dam was used for isolation. Before the replacement of composite restorations, enamel edges were etched according to selective etching method. Then universal adhesive system was applied. Composite resin was applied to the cavity in 2 mm layers by incramental technique. Glass carbomer was placed with bulk technique by applying finger pressure with surface covering. Composite restorations were polymerized with LED light curing unit. Glass carbomer restorations were cured its own special curing unit. Restorations were evaluated with modified USPHS criteria at the end of the first week, 6 months and 12 months. Data were analyzed using Fisher's Exact Chi-Square test, Fisher Freeman Halton Test and Continuity (Yates) Correction. Wilcoxon sign test was used for intra-group comparisons of the parameters. Statistically significance was evaluated at p <0.05.

ELIGIBILITY:
Inclusion Criteria:

1. 20-25 years of age
2. No systemic diseases
3. Presence of molar / premolar teeth with occlusal and / or interface caries
4. Lack of parafunctional habits such as clenching and grinding of teeth
5. Lack of cooperation problems
6. Accepted regular visits -

Exclusion Criteria:

* 1-Any endodontic treatment or withdrawal indications (abscess, swelling and fistula complaints, palpation and percussion pain, spontaneous or night pain) 2- Teeth with congenital developmental defect 3- Teeth with pathological mobility 4- Teeth which do not have normal occlusion due to skeletal or pathological reasons 5- Lack of contact or opposite teeth

Ages: 25 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2017-09-09 (Actual); Primary Completion 2017-09-16 (Actual); Study Completion 2018-09-10 (Actual)

PRIMARY OUTCOMES:
Evaluation of criterias | 1 week
  In this clinical study, the restorations were evaluated.Restorations were scored. using the terms Alpha, Bravo and Charlie.Alpha was used for restorations that were considered clinically successful; Bravo was used for the restorations with several deficiencies but requiring no replacement; and Charlie was used for the clinically unacceptable restorations where the restoration had to be replaced.End of the one-week there was no significant differences between restorative materials for all evaluation criterias, were mentioned in summary.

SECONDARY OUTCOMES:
Evaluation of criterias | 6-months
  In this clinical study, the restorations were evaluated.Restorations were scored using the terms Alpha, Bravo and Charlie.Alpha was used for restorations that were considered clinically successful; Bravo was used for the restorations with several deficiencies but requiring no replacement; and Charlie was used for the clinically unacceptable restorations where the restoration had to be replaced.2. When the restorations made using glass carbomer filling materials were evaluated in terms of anatomic form, retention, and marginal adaptation, restorations with Charlie score in the 6-months

OTHER OUTCOMES:
Evaluations of criterias | 12-months
  In this clinical study, the restorations were evaluated.Restorations were scored using the terms Alpha, Bravo and Charlie.Alpha was used for restorations that were considered clinically successful; Bravo was used for the restorations with several deficiencies but requiring no replacement; and Charlie was used for the clinically unacceptable restorations where the restoration had to be replaced.2. When the restorations made using glass carbomer filling materials were evaluated in terms of anatomic form, retention, and marginal adaptation, restorations with Charlie score in the 12-months.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Buket Kaynar, Dr, Principal Investigator — Bezmialem Vakif University
Locations (1):
- Bezmialem vakif university, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 12 months